CLINICAL TRIAL: NCT01498796
Title: KITS Study -Ketorolac In Tonsillectomy Surgery: a Double Blinded, Randomized Clinical Trial
Acronym: KITS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI no longer at institution
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: Pro00002357
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Recurrent Acute Tonsillitis
MeSH Terms: interventions — Ketorolac; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketorolac (Experimental)
  Interventions: Drug: Ketorolac
- Placebo (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Ketorolac
  Arms: Ketorolac
Drug: Normal Saline
  Arms: Placebo

SUMMARY:
Our group wishes to test the novel hypothesis that intraoperative use of ketorolac in pediatric patients undergoing tonsillectomy reduces post-operative nausea and vomiting, postoperative pain scores, subsequent narcotic use, and length of hospital stay without adversely affecting post-operative bleed risk, when compared to placebo, in a double-blind, randomized controlled trial.

DETAILED DESCRIPTION:
Intraoperative analgesia has a tremendous theoretical potential to decrease postoperative pain, and thus narcotic requirement and length of subsequent hospital stay. There is indeed a dearth of evidence with respect to the clinical effectiveness of such analgesia. Tonsillectomy lends itself particularly well to the use of intraoperative analgesia; post-operative pain scores are high, and the majority of recipients are pediatric patients-a population in which minimization of post-operative narcotic use is a priority.

The effectiveness of intraoperative analgesia for the preemptive management of postoperative pain, nausea and vomiting in tonsillectomy remains controversial. Pre-emptive analgesia was first conceptualized in 1983, with Woolf's work on a postulated central component of postinjury pain hypersensitivity. Tissue injury is typified by post-stimulus sensory disturbances that give rise to continuing pain, a hypersensitivity to further noxious stimuli, as well as pain in response to otherwise innocuous stimuli. These features are attributable to both a reduction in the threshold of skin nociceptors, as well as an increase in the excitability of the central nervous system (CNS) to noxious stimuli. Much experimental data has shown pre-injury analgesia as being superior to post-injury analgesia in terms of minimizing subsequent CNS excitability.

Clinically, the effectiveness of such analgesia has shown to be highly variable with respect to anatomical area, surgical type, as well as analgesic used and its route of administration. A Meta-analysis by Cliff et al. reviewed 66 studies with respect to the primary outcomes of pain intensity scores, supplemental analgesic consumption, and time to first analgesic consumption, and demonstrated that preemptive administration of NSAIDs was superior to that of epidural analgesia, local anesthetic wound infiltration, systemic NMDA receptor antagonists, and systemic opiods.

Ketorolac tromethamine (Toradol) is a parenteral, nonsteroidal anti-inflammatory drug that has been used extensively to provide postoperative analgesia. In a prospective, randomized double-blind study of 57 children undergoing outpatient adenotonsillectomy, Keidan et al. found ketorolac to be comparable to fentanyl in terms of both post-operative nausea and vomiting and pain scores. One study showed that intraoperative ketorolac (60 mg IV) with fentanyl (2 micrograms/kg IV), compared to fentanyl and placebo, administered at the induction of anesthesia resulted in significant opioid sparing, decreased pain scores, lower incidence of nausea and vomiting and earlier discharge compared to fentanyl and placebo in patients undergoing diagnostic laparoscopy.

There is a theoretical risk of post-operative bleeding with use of Toradol, on account of its inhibition of platelet aggregation and prolonging of bleeding time. However, in a meta-analysis of 13 trials comprising 955 children undergoing tonsillectomy, Cardwell et al. found that postoperative NSAIDs did not significantly alter number of perioperative bleeding events requiring surgical intervention. At present, it is common practice by some clinicians at the Stollery Children's hospital for pediatric patients who are undergoing standard electrocautery adenotonsillectomy to receive intraoperative ketorolac. Its role in improving post-operative pain and possible risk of increasing post-operative bleeding remains controversial.

i Woolf CJ: Evidence for a central component of post-injury pain hypersensitivity. Nature 1983; 308: 386-8

ii Coderre TJ, Catz J, Vaccarino AL, Melzack R: Contribution of central neutoplasticity to pathological pain: Review of clinical and experimental evidence. Pain 1993; 52: 259-85

iii Aida S, Baba H, Yamakura T, MD, Taga K, Fukuda S, Shimoji K: The Effectiveness of Preemptive Analgesia Varies According to the Type of Surgery: A Randomized, Double-Blind Study. Anesth Analg 1999;89: 711 ivOng CKS, Lirk P, Seymour RA, Jenkins BJ: The Efficacy of Preemptive Analgesia for Acute Postoperative Pain Management: A Meta-Analysis. Anesth Analg 2005;100:757-773

v Keidan I, Zaslansky R, Eviatar E, Segal S, Sarfaty SM. Intraoperative ketorolac is an effective substitute for fentanyl in children undergoing outpatient adenotonsillectomy.

Paediatric Anaesthesia. 14(4):318-23, 2004 Apr.

vi Green CR, Pandit SK, Levy L, Kothary SP, Tait AR, Schork MA Intraoperative ketorolac has an opioid-sparing effect in women after diagnostic laparoscopy but not after laparoscopic tubal ligation. Anesthesia & Analgesia. 82(4):732-7, 1996 Apr.

vii Cardwell M, Siviter G, Smith A Non-steroidal anti-inflammatory drugs and perioperative bleeding in paediatric tonsillectomy. Cochrane Database of Systematic Reviews. Issue: 2 Article: CD003591, 2005

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3yrs-15yrs who will undergo tonsillectomy or adeno-tonsillectomy for sleep disordered breathing confirmed by oximetry

Exclusion Criteria:

* Severe Obstructive Sleep Apnea
* Co-morbid disease precluding use of NSAIDS or Narcotics
* Language/developmental/social inability to assess pain scores

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pain post-tonsillectomy | post-operative
  pain post-tonsillectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada